CLINICAL TRIAL: NCT07238595
Title: Relationship Between Cervical Pain, Functional Fitness, and Kinesiophobia According to Cervical Proprioceptive Awareness Level in the Healthy Elderly
Brief Title: Relationship Between Cervical Pain According to Cervical Proprioceptive Awareness Level in the Healthy Elderly
Status: Enrolling by invitation | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Melik AVCI, MSc student, physiotherapist, Suleyman Demirel University
Other Study IDs: SuleymanDU
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Elderly (People Aged 65 or More)
Keywords: Elderly; Cervical proprioception; Cervical pain; Functional Fitness; Kinesiophobia
MeSH Terms: conditions — Neck Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- older adults with high cervical proprioceptive awareness: In this study, several standardized assessments will be administered to evaluate different physical and cognitive parameters of older adults. Cognitive functions will be assessed using the Standardized Mini-Mental Test (SMMT). Cervical proprioceptive awareness will be measured with the Cervical Joint Position Error Test (CJPE), which uses a laser-guided system to assess joint position sense. Pain intensity, quality, and its impact on daily living activities will be evaluated with the Geriatric Pain Scale (GPS). Physical fitness parameters such as strength, balance, flexibility, and agility will be measured through the Senior Fitness Test (SFT), which includes multiple functional subtests. Finally, fear of movement related to pain will be assessed using the Tampa Scale of Kinesiophobia (TSK). All assessments will be conducted by a physiotherapist under standardized testing conditions.
  Interventions: Other: Cervical Joint Position Error Test (CJPE)
- older adults with low cervical proprioceptive awareness: In this study, several standardized assessments will be administered to evaluate different physical and cognitive parameters of older adults. Cognitive functions will be assessed using the Standardized Mini-Mental Test (SMMT). Cervical proprioceptive awareness will be measured with the Cervical Joint Position Error Test (CJPE), which uses a laser-guided system to assess joint position sense. Pain intensity, quality, and its impact on daily living activities will be evaluated with the Geriatric Pain Scale (GPS). Physical fitness parameters such as strength, balance, flexibility, and agility will be measured through the Senior Fitness Test (SFT), which includes multiple functional subtests. Finally, fear of movement related to pain will be assessed using the Tampa Scale of Kinesiophobia (TSK). All assessments will be conducted by a physiotherapist under standardized testing conditions.
  Interventions: Other: Cervical Joint Position Error Test (CJPE)

INTERVENTIONS:
Other: Cervical Joint Position Error Test (CJPE) — The Cervical Joint Position Error Test (CJPE) is a clinical assessment used to evaluate cervical proprioceptive awareness by measuring how accurately a person can reposition their head to a neutral position after active neck movements. During the test, a laser pointer attached to the participant's head projects onto a target, and the difference between the starting and returning points is recorded. Smaller errors indicate better proprioceptive control and joint position sense in the cervical region.

SUMMARY:
Aging is a progressive and irreversible process characterized by changes occurring at the cellular level, in organs and systems. Kinesiophobia in older adults is defined as a condition in which an individual is unable to perform movement due to fear of pain or injury. Studies have shown that with increasing age, kinesiophobia also increases, leading to a decrease in physical activity. In older individuals with chronic neck pain, significant relationships have been found between kinesiophobia, proprioceptive position error (JPE), and functional performance. Kinesiophobia is strongly associated with pain intensity and stands out as an important factor that negatively affects proprioceptive perception and functional performance, particularly in neck extension and rotation movements (for example, handgrip strength).

In summary, decreased proprioception in older adults may lead to reduced functional fitness and increased kinesiophobia. This may cause the individual to avoid movement, leading to a vicious cycle in which proprioceptive sense and functional capacity further deteriorate. The aim of this study is to examine the relationship between cervical pain, functional fitness, and kinesiophobia according to the level of cervical proprioceptive awareness in healthy older adults.At least 60 individuals with high proprioceptive awareness and 60 individuals with low cervical proprioceptive awareness will be included in the study. First, a sociodemographic data form will be completed. The Standardized Mini-Mental Test will be administered to assess the participants' cognitive functions. Then, the Cervical Joint Position Error Test will be used to evaluate the sense of position in the neck region. The Geriatric Pain Scale will be applied to assess the participants' pain levels; this scale is used to evaluate the intensity, quality, and impact of pain on daily living activities in older adults. Finally, the Tampa Scale of Kinesiophobia will be used to assess fear of movement. Participants will complete the 17-item self-report questionnaire under the supervision of a physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65
* mini mental test score ≥ 24
* Being independent in physical functions
* Being able to read and write in Turkish
* Consent to participate in the study

Exclusion Criteria:

* Having a history of cervical surgery
* Experiencing cervical trauma within the past month
* Having neurological diseases such as dementia or Alzheimer's
* Having cognitive impairment
* Having other musculoskeletal problems that may affect the cervical region, such as impingement, thoracic outlet syndrome, or scoliosis
* Using assistive devices for walking and/or standing
* Using more than four medications per day
* Having vision problems that are not corrected despite visual aids
* Having specific pathological conditions such as malignancy, fractures, or systemic rheumatoid disease
* Having a diagnosed psychiatric disorder
* Receiving medical treatment that may affect balance and posture

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults over 65 years with high cervical proprioceptive awareness in the study group
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11-29 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Cervical Joint Position Error Test | one day
  The Cervical Joint Position Error Test is a clinical assessment used to evaluate cervical proprioceptive awareness by measuring how accurately a person can reposition their head to a neutral position after active neck movements. During the test, a laser pointer attached to the participant's head projects onto a target, and the difference between the starting and returning points is recorded. Smaller errors indicate better proprioceptive control and joint position sense in the cervical region.
Cervical Joint Position Error Test (CJPE) | 1 day
  The Cervical Joint Position Error Test (CJPE) is a clinical assessment used to evaluate cervical proprioceptive awareness by measuring how accurately a person can reposition their head to a neutral position after active neck movements. During the test, a laser pointer attached to the participant's head projects onto a target, and the difference between the starting and returning points is recorded. Smaller errors indicate better proprioceptive control and joint position sense in the cervical region.

SECONDARY OUTCOMES:
Standardized Mini-Mental Test (SMMT) | one day
  The Standardized Mini-Mental Test (SMMT) is a brief cognitive assessment tool used to evaluate various aspects of mental function in older adults. It measures domains such as orientation, attention, memory, language, and visuospatial abilities, providing an overall score out of 30 points. Higher scores indicate normal cognitive function, while lower scores suggest different levels of cognitive impairment. The test takes approximately 10 minutes to administer and is widely used for screening cognitive status, particularly in identifying mild to severe cognitive decline.
Geriatric Pain Scale | one day
  The Geriatric Pain Scale (GPS) is an assessment tool designed to evaluate pain intensity, quality, and its impact on daily living activities in older adults. It consists of multiple items that explore the frequency, duration, and nature of pain, as well as movement limitations and pain management strategies. The scale helps clinicians understand the overall pain experience of elderly individuals and its effect on their functional abilities. It is easy to administer, typically taking about 5-10 minutes, and provides valuable insight for developing appropriate pain management interventions.
Senior Fitness Test (SFT) | one day
  The Senior Fitness Test (SFT) is a comprehensive assessment used to evaluate the physical fitness of older adults. It measures key components such as muscle strength, flexibility, balance, agility, and cardiovascular endurance through a series of functional subtests, including chair stands, arm curls, walking tests, and reach or flexibility tasks. The SFT provides objective information about an individual's functional abilities, helping to identify areas that may benefit from targeted exercise or rehabilitation programs.
Tampa Scale of Kinesiophobia | one day
  The Tampa Scale of Kinesiophobia (TSK) is a self-report questionnaire designed to assess fear of movement or reinjury due to pain. It consists of 17 items rated on a 4-point Likert scale, measuring the degree to which individuals avoid physical activity because of pain-related anxiety. The TSK helps clinicians identify patients at risk of activity limitation and guides interventions to reduce fear-avoidance behaviors, ultimately supporting improved functional outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Melik AVCI, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alahmari KA, Reddy RS, Silvian P, Ahmad I, Nagaraj V, Mahtab M. Influence of chronic neck pain on cervical joint position error (JPE): Comparison between young and elderly subjects. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1265-1271. doi: 10.3233/BMR-169630. PMID 28800305
- See also: Proprioceptive sensibility in the elderly: degeneration, functional consequences and plastic-adaptive processes — https://pubmed.ncbi.nlm.nih.gov/28800305/